CLINICAL TRIAL: NCT00251836
Title: Prospective Evaluation of Adrenal Function After Living Donor Nephrectomy With or Without Ligation of the Adrenal Vein
Brief Title: Adrenal Function After Living Kidney Donation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: StV 34-2005; RAB-F-02-0046
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Addison Disease; Hypoaldosteronism
Keywords: Kidney donation; Organ Donation; Vascular anatomy; Adrenal Insufficiency
MeSH Terms: conditions — Addison Disease; Hypoaldosteronism; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left-sided donor nephrectomy: Left-sided laparoscopic hand-assisted donor nephrectomy
  Interventions: Procedure: Laparoscopic hand-assisted donor nephrectomy
- Right-sided donor nephrectomy: Right-sided laparoscopic hand-assisted donor nephrectomy
  Interventions: Procedure: Laparoscopic hand-assisted donor nephrectomy

INTERVENTIONS:
Procedure: Laparoscopic hand-assisted donor nephrectomy

SUMMARY:
The success of kidney transplantation is hampered by the shortage of organs. One attractive strategy is the use of kidneys from living donors. During the donor operation the kidney artery, kidney vein and ureter have to be interrupted as far as possible from the kidney to have sufficient length for the reconnection of these structures in the transplant operation.

An adrenal gland is situated at the upper pole of each kidney. While the arterial supply is accomplished by many small vessels, the venous drainage is only through one vein. On the right side the adrenal vein empties directly into the inferior vena cava (the large vessel transporting blood from the lower body to the heart). In contrast, on the left side the adrenal vein empties into the kidney vein, which in turn drains to the inferior vana cava. Due to these anatomical differences a left-sided removal of a kidney always necessitates an interruption of the left adrenal vein, while a right-sided kidney removal does not.

As the venous drainage of the left adrenal gland is closed during living kidney donation, the gland is most likely functionally impaired. This can be compared to a right-sided kidney donation, where the adrenal vein is left intact. These comparisons are performed by adrenal function tests before, one week after and one month after kidney donation. These function tests consist of blood values drawn after stimulation with a hormone drug.

DETAILED DESCRIPTION:
Due the lack of suitable donor organs a large proportion of kidney transplantations is now performed from living donors. In the year 2002 the number of living donors surpassed the number of cadaveric donors in Switzerland (Swisstransplant, Swiss Transplant Society 2005). Kidney grafts from living donors have superior long-term outcome (Hariharan S, N Engl J Med 2000). At the University Hospital Zurich 28 of the 84 kidney transplantations performed in the year 2004 were from living donors.

During living donor nephrectomy the renal artery and renal vein are transected as far away from the kidney as possible, to ensure an adequate vessel length for the subsequent transplantation procedure. The arterial supply of the adrenal glands is accomplished by several small vessels (ca. 5-15), while the venous drainage is usually dependent on a single vein. While the right-sided adrenal vein drains directly into the inferior vena cava (IVC), the left-sided adrenal vein drains into the renal vein. Variants are relatively rare and occur in 5% of cases (Sebe P, Surg Radiol Anat 2002). Therefore, during donor nephrectomy of the left kidney the adrenal vein is transected, while this is not necessary on the right side.

The question addressed in this clinical trial is whether left-sided donor nephrectomy affects the left adrenal gland. This might be compensated immediately by the contralateral gland or it might lead to a measurable functional adrenal deficit. Such an adrenal insufficiency could be detrimental to the immediate postoperative course. The intermediate-term outcome of the adrenal glands is also of interest, as an impairment of the left adrenal gland will lead to a hypertrophy of the contralateral gland.

Few scientific publications have addressed these questions. There are case reports of acute intra- and postoperative adrenal insufficiency in patients undergoing nephrectomy with adrenalectomy (Cassinello Ogea C, Rev Esp Anestesiol Reanim 2002, Henrich WL, Urology 1976, Messiant F, Ann Fr Anesth Reanim 1993, Safir MH, Geriatr Nephrol Urol 1998). A small prospective study in patients undergoing radical nephrectomy (including adrenalectomy) did not find signs of adrenal insufficiency (Bischoff P, Anaesthesist 1997). However a subgroup analysis of a newer study demonstrated adrenal insufficiency in radical versus adrenal-sparing nephrectomy (Yokoyama H, BJU Int 2005).

The study hypothesis is that left-sided donor nephrectomy (i.e. with transaction of the adrenal vein) is deleterious to the left adrenal gland and causes a measurable transient adrenal insufficiency after the operation. The primary study endpoint is the assessment of adrenal function after donor nephrectomy. This is done by an ACTH stimulation test, performed at baseline, in the first week after the operation and 4 weeks after the operation. Comparisons are performed between baseline and postoperative values, as well as between left-sided kidney donors (n=20) and right-sided kidney donors (n=10). A secondary study endpoint is to assess the morphological response of both adrenal glands after donor nephrectomy. To this end MRI and volumetry of the adrenal glands is performed at the same time points, with the hypothesis that left-sided nephrectomy will lead to an involution of the left adrenal followed by hypertrophy of the right adrenal.

ELIGIBILITY:
Inclusion Criteria:

* Eligible kidney donor (meeting institutional selection criteria)
* Informed consent for study participation

Exclusion Criteria:

* Treatment with glucocorticoids
* Preexisting diseases of adrenal function (hypercortisolism, hyperaldosteronism, adrenal insufficiency)
* Inability to undergo MRI examination (metal implants, etc.)
* Inability to understand the study information and to give informed consent (in German)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible living donors were considered for participation in the study unless exclusion criteria were present: active corticoid medication, known adrenal disease such as hypercortisolism, hyperaldosteronism or adrenal insufficiency, or the presence of metallic implants precluding MRI investigation. All living kidney donor candidates underwent a standard somatic and psychological eligibility testing during a brief hospitalization in accordance with the Swiss Transplantation Act and the guidelines of the Swiss Academy of Medical Sciences.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Plasma cortisol response to low-dose ACTH stimulation | Pre-operative, day 1 and day 28 after kidney donation
  Low-dose ACTH1-24 stimulation test was conducted by drawing blood at 8 am, then injecting 1 Ig of Synacthen intravenously and drawing further blood samples after 30, 60, and 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weber, MD, Principal Investigator — Dept. of Visceral and Transplantation Surgery, University Hospital Zurich
Locations (1):
- Dept. of Visceral and Transplantation Surgery, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hariharan S, Johnson CP, Bresnahan BA, Taranto SE, McIntosh MJ, Stablein D. Improved graft survival after renal transplantation in the United States, 1988 to 1996. N Engl J Med. 2000 Mar 2;342(9):605-12. doi: 10.1056/NEJM200003023420901. PMID 10699159
- [Background] Sebe P, Peyromaure M, Raynaud A, Delmas V. Anatomical variations in the drainage of the principal adrenal veins: the results of 88 venograms. Surg Radiol Anat. 2002 Aug-Sep;24(3-4):222-5. doi: 10.1007/s00276-002-0021-x. Epub 2002 Jun 13. PMID 12375078
- [Background] Cassinello Ogea C, Giron Nombiela JA, Ruiz Tramazaygues J, Izquierdo Villarroya B, Sanchez Tirado JA, Almajano Dominguez RM, Oro Fraile J. [Severe perioperative hypotension after nephrectomy with adrenalectomy]. Rev Esp Anestesiol Reanim. 2002 Apr;49(4):213-7. Spanish. PMID 14606383
- [Background] Henrich WL, Goldberg J, Lucas M, Gabow P. Adrenal insufficiency after unilateral radical nephrectomy. Urology. 1976 Dec;8(6):584-5. doi: 10.1016/0090-4295(76)90525-2. PMID 997054
- [Background] Messiant F, Duverger D, Verheyde I, Declerck N, Pruvot FR, Scherpereel P. [Postoperative acute adrenal insufficiency]. Ann Fr Anesth Reanim. 1993;12(6):594-7. doi: 10.1016/s0750-7658(05)80629-x. French. PMID 8017676
- [Background] Safir MH, Smith N, Hansen L, Kozlowski JM. Acute adrenal insufficiency following unilateral radical nephrectomy: a case report. Geriatr Nephrol Urol. 1998;8(2):101-2. doi: 10.1023/a:1008305627588. PMID 9893218
- [Background] Bischoff P, Noldus J, Harksen J, Bause HW. [The necessity for perioperative cortisol substitution. Spontaneous and stimulated ACTH and cortisol secretion during unilateral adrenalectomy for renal cell carcinoma]. Anaesthesist. 1997 Apr;46(4):303-8. doi: 10.1007/s001010050405. German. PMID 9229984
- [Background] Yokoyama H, Tanaka M. Incidence of adrenal involvement and assessing adrenal function in patients with renal cell carcinoma: is ipsilateral adrenalectomy indispensable during radical nephrectomy? BJU Int. 2005 Mar;95(4):526-9. doi: 10.1111/j.1464-410X.2005.05332.x. PMID 15705073